CLINICAL TRIAL: NCT04439747
Title: Develop and Implement Methods for Diagnostic and Treatment of Hormonal Disorders in Patients With Chronic Kidney Disease
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Belarusian State Medical University (Other)
Responsible Party: Principal Investigator, Tatiana Mokhort, Professor, MD, Head of Endocrinology Department, Belarusian State Medical University
Other Study IDs: 20180438
Record Dates: First submitted 2020-06-17; First posted 2020-06-19 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Hyperprolactinemia; Thyroid Dysfunction; Bone Diseases, Metabolic; Chronic Kidney Diseases
Keywords: hormonal alterations, RRT, CKD, kidney transplantation
MeSH Terms: conditions — Hyperprolactinemia; Bone Diseases, Metabolic; Renal Insufficiency, Chronic | interventions — High-Energy Shock Waves; Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control: Ultrasound examination of the thyroid gland and parathyroid glands, osteodensitometry (DXA), biochemical analysis, general blood count, neutrophil- gelatinase assosiated lipocalin-2 (NGAL), adiponectin, urine albumin / creatinine ratio, hormonal tests (TSH, free T4 and T3, total T4 and T3, Tg, antibodies to thyroid peroxidase (Ab-TPO), Ab--R-TSH, Ab-Tg, parathyroid hormone (PTH), vitamin D, osteocalcin, b-cross-laps, prolactin)
  Interventions: Other: Ultrasound, DXA, hormonal tests
- CKD 1-2: Ultrasound examination of the thyroid gland and parathyroid glands, osteodensitometry (DXA), biochemical analysis, general blood count, NGAL, adiponectin, urine albumin / creatinine ratio, hormonal tests (TSH, free T4 and T3, total T4 and T3, Tg, Ab-TPO, Ab--R-TSH, Ab-Tg, PTH, vitamin D, osteocalcin, b-cross-laps, prolactin)
  Interventions: Other: Ultrasound, DXA, hormonal tests
- CKD 3-5: Ultrasound examination of the thyroid gland and parathyroid glands, osteodensitometry (DXA), biochemical analysis, general blood count, NGAL, adiponectin, urine albumin / creatinine ratio, hormonal tests (TSH, free T4 and T3, total T4 and T3, Tg, Ab-TPO, Ab--R-TSH, Ab-Tg, PTH, vitamin D, osteocalcin, b-cross-laps,prolactin)
  Interventions: Other: Ultrasound, DXA, hormonal tests

INTERVENTIONS:
Other: Ultrasound, DXA, hormonal tests — Diagnostic tests in selected groups with investigation of revealed hormonal disorders

SUMMARY:
Methods of diagnostic and treatment of hormonal disorders in patients with chronic kidney disease (CKD) will be developed and implemented in real clinical practice. As a result of the project, new scientific data will be obtained on the relationship of hyperprolactinemia and impaired functioning of the pituitary-gonadal axis, changes in functioning of the renin-angiotensin-aldosterone system will be revealed, and the characteristics of the thyroid and parathyroid status in patients with CKD will be determined, including receiving renal replacement therapy (RRT) and after kidney transplantation, which will improve the efficiency of diagnosis and treatment of hormonal disorders in the early stages of the disease, reduce the direct financial costs of the diagnostic and treatment process primarily due to the optimization of hormonal studies and treatment of the revealed disorders, as well as will prevent the progression of CKD and the severity of the condition of this category of patients due to the development of hormonal dysfunctions.

DETAILED DESCRIPTION:
1. Assessment of prevalence, clinical manifestations and pathological significance in a cohort of patients with CKD:

   * hyperprolactinemia, hormonal disorders of a pituitary -gonad axis ;
   * disorders of renin-angiotensin-aldosterone system;
   * pathology of the thyroid and parathyroid glands.
2. Analysis of CKD impact on the development of structural changes in the thyroid gland and parathyroid glands according to the results of ultrasound examination.
3. Assessment of relationship of hormonal dysfunctions in patients with CKD and adipocytokines, markers of renal impairment.
4. To study the effect of renal replacement therapy on thyroid hormones clearance .
5. Investigate hormonal status in patients with CKD after kidney transplantation.

ELIGIBILITY:
Inclusion Criteria:

* patients at CKD 1-5, including renal replacement therapy and renal transplantation

Exclusion Criteria:

* patients with impaired thyroid function before the onset of CKD;
* pregnant women;
* patients with acute diseases;
* patients in the acute phase of comorbid chronic diseases;
* patients in the acute period of myocardial infarction, after acute cerebrovascular accident;
* patients with mental illness;
* patients undergoing treatment for various cancer types.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients of nephrology departments in Minsk City hospitals and endocrinology department of Minsk Endocrinology Dispensary from which 2 groups will be selected , healthy volunteers of Minsk as control group
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Hormanal changes in patients with CKD | Baseline
  Deviations from reference interval ranges of prolactin, thyroid hormones, PTH and vitamin D and its associations with renal impairment markers

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Mokhort, Prof, Study Chair — Head of Endocrinology Department
Locations (1):
- Belarusian State Medical University Endocrinology Department, Minsk, Belarus

IPD SHARING:
Plan to Share IPD: No